CLINICAL TRIAL: NCT04171505
Title: Retrospective Cohort Study to Analyze Whether Prophylactic Vaccination Against HPV Can Reduce the Risk of Recurrence in Women Who Have Received an Excisional Therapy for HSIL / CIN2-3. Recurrence is Defined as the Detection of Infection by the Same HPV Genotype for at Least 6-12 Months (Persistent Infection), and / or Cytological Alteration and / or Cervical and / or Vaginal Histological Lesion of Any Grade (SIL / CIN / VaIN) in Patients With Negative Cotest in the First Post Control.
Brief Title: Retrospective Cohort Study of the Effectiveness of the Prophylactic Vaccine Against the Human Papilloma Virus in the Prevention of Recurrence in Women Who Have Received an Excisional Therapy by HSIL / CIN.
Acronym: VENUS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital San Carlos, Madrid (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, ANDREA CASAJUANA, PLUVIO CORONADO MARTÍN, Hospital San Carlos, Madrid
Other Study IDs: ISM-190623
Record Dates: First submitted 2019-11-19; First posted 2019-11-21 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Cervix, Dysplasia; HPV Infection; HPV Vaccine; Cervix Lesion
MeSH Terms: conditions — Uterine Cervical Dysplasia; Papillomavirus Infections | interventions — Papillomavirus Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- vaccinated women: * Women older than 18 years who received excisional therapy due to HSIL /CIN injury confirmed histologically.
  * Women who sign informed consent.
  * Patients with negative results in the first post-surgery control.
  * Patients who have received HPV vaccination and provide vaccination card.
  Interventions: Drug: HPV vaccine
- non vaccinated woman: * Women older than 18 years who received excisional therapy due to HSIL /CIN injury confirmed histologically.
  * Women who sign informed consent.
  * Patients with negative results in the first post-surgery control.
  * Patients who have NOT received HPV vaccination and provide vaccination card.

INTERVENTIONS:
Drug: HPV vaccine — . Patients diagnosed with HSIL / CIN 2+ who met the inclusion criteria were submitted to cervical conization and subsequently enrolled in the study after signing the informed consent, approved by ethics commission.
  We will take into account the date of administration of the first dose of vaccine. The types of vaccines administered can be: Bivalent vaccine (includes genotypes 16/18), Tetravalent (includeds genotypes 6, 11, 16 and 18) both funded in the region in different years, or not funded (Nonavalent vaccine; includes genotypes: 6, 11, 16, 18, 31, 33, 45, 52 and 58). To define the time of vaccination around the conization date, the administration of the first dose of vaccine will be taken into account.
  Groups: vaccinated women

SUMMARY:
A retrospective cohort study of women treated by excisional therapy due to HSIL/ CIN at Clínico San Carlos Hospital between 2012-2018. The effectiveness of prophylactic vaccination against HPV in women treated for HPV-related disease will be evaluated. For this purpose, the percentage of cervical lesion recurrence among a group of treated and vaccinated women against HPV between the years 2015-2018 will be compared with a control group of treated and non-vaccinated women against HPV since 2012-2015.

It will be an essential requirement that the patient provide a vaccination card from their health center where there is proof of their immunization status and date of administration.

Inclusion criteria:

* Women older than 18 years who received excisional therapy due to HSIL /CIN injury confirmed histologically.
* Women who sign informed consent.
* Patients with negative results in the first post-surgery control.
* Patients who have received HPV vaccination and provide vaccination card.

Exclusion criteria:

* Women who do not wish or cannot give their informed consent and / or do not comply with the requirements of the study.
* Patients treated by an indication other than HSIL/CIN.
* Patients under immunosuppression conditions.

DETAILED DESCRIPTION:
A retrospective cohort study of women treated by excisional therapy due to HSIL/ CIN at Clínico San Carlos Hospital (Madrid) between 2012-2018. The effectiveness of prophylactic vaccination against HPV in women treated for HPV-linked disease will be evaluated. For this purpose, the percentage of lesional recurrence among a group of treated and vaccinated women against HPV between the years 2015-2018 will be compared with a control group of treated and non-vaccinated women against HPV since 2012-2015. The data will be obtained through the review of clinical records.

Our protocol is explained above:

HPV detection method:

The detection of HPV is performed on a liquid basis by means of the CLARK PAPILOMAVIRUS HUMAN test that detects the presence of the HPV virus (6, 11, 16, 18, 26, 31, 33, 35, 39, 40, 42, 43, 44, 45, 51, 52, 53, 54, 56, 58, 59, 61, 62, 66, 68, 70, 71.72, 73, 81, 82, 83, 84, 85 and 89). The test has a diagnostic sensitivity of 98.2% and a diagnostic specificity of 100% and analytical specificity: 100%. The analytical sensitivity of this test is 100% when the number of copies is 1,000 or 10,000 depending on the type of HPV. The Laboratory has carried out external quality control of the SEAP.

Pre-surgical evaluation:

Those patients with an abnormal cytological result and / or positive HPV tests were referred to the PTGI consultations of Clínico San Carlos Hospital for evaluation according to the Cervical Cancer Prevention Guidelines issued by the Spanish Association of Cervical Pathology and Colposcopy (AEPCC) in 2006 and 2014. These patients underwent colposcopy with biopsy if necessary +/- determination of HPV. Patients diagnosed with HSIL / CIN 2+ who met the inclusion criteria were submitted to cervical conization and subsequently enrolled in the study after signing the informed consent, approved by ethics commission.

We will take into account the date of administration of the first dose of vaccine. The types of vaccines administered can be: Bivalent vaccine (includes genotypes 16/18), Tetravalent (includeds genotypes 6, 11, 16 and 18) both funded in the region in different years, or not funded (Nonavalent vaccine; includes genotypes: 6, 11, 16, 18, 31, 33, 45, 52 and 58). To define the time of vaccination around the conization date, the administration of the first dose of vaccine will be taken into account.

Surgical treatment:

Excisional therapy was performed in the operating room on a scheduled basis under local analgesia and sedation. After infiltration with local anesthetic and vasoconstrictor in the 4 quadrants of the cervix, excisional therapy with diathermic loop is performed under colposcopy control, obtaining the piece in a single specimen. The piece is oriented with a long thread at 12:00 h, it is introduced in formaldehyde and send to pathological anatomy for deferred study. In all cases, immediate endocervical curettage post-treatment was performed.

Clinical follow-up:

The first revision is made 30 days after surgery where patient is informed of histological results and the date on first control post-treatment based on the diagnosis.

Following the protocol of the AEPCC, in case of non-involvement of margins and negative endocervical curettage, the patient comes after 6 months from the intervention to perform the first post-surgery control with co-test. In case of positive endocervical curettage or margin involvement, the first post-surgery control will be performed at 4 months with cotest + endocervical study and colposcopy. Persistent disease is defined as the presence of cytological alteration and / or HPV infection in the first post control performed at 4-6 months after excisional therapy. These patients are excluded from the study, since only those in which both tests are negative will be included.

Subsequently, a new co-test was performed at 12 months, 24 months and 36 months after the first post-surgery control. After 3 years of negative testing, the patient is returned to the current cervical cancer-screening program.

ELIGIBILITY:
Inclusion Criteria:

* Women older than 18 years who received excisional therapy due to HSIL /CIN injury confirmed histologically.
* Women who sign informed consent.
* Patients with negative results in the first post-surgery control.
* Patients who have received HPV vaccination and provide vaccination card.

Exclusion Criteria:

* Women who do not wish or cannot give their informed consent and / or do not comply with the requirements of the study.
* Patients treated by an indication other than HSIL/CIN.
* Patients under immunosuppression conditions.

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women treated by excisional therapy due to HSIL/ CIN at Clínico San Carlos Hospital between 2012-2018
Sampling Method: Non-Probability Sample
Enrollment: 508 (Estimated)
Dates: Start 2019-11-04 (Actual); Primary Completion 2019-11-04 (Actual); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Recurrence | 2 years
  defined as the existence of persistent HPV infection and / or presence of cytological abnormality and / or presence of SIL / CIN / VaIN of any grade.

SECONDARY OUTCOMES:
Age, type of virus, degree of injury, variables related to demographic and histological data of the patient, date of 1st dose of vaccine. | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinico San Carlos, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kang WD, Choi HS, Kim SM. Is vaccination with quadrivalent HPV vaccine after loop electrosurgical excision procedure effective in preventing recurrence in patients with high-grade cervical intraepithelial neoplasia (CIN2-3)? Gynecol Oncol. 2013 Aug;130(2):264-8. doi: 10.1016/j.ygyno.2013.04.050. Epub 2013 Apr 26. PMID 23623831
- [Result] FUTURE II Study Group. Quadrivalent vaccine against human papillomavirus to prevent high-grade cervical lesions. N Engl J Med. 2007 May 10;356(19):1915-27. doi: 10.1056/NEJMoa061741. PMID 17494925
- [Result] Ghelardi A, Parazzini F, Martella F, Pieralli A, Bay P, Tonetti A, Svelato A, Bertacca G, Lombardi S, Joura EA. SPERANZA project: HPV vaccination after treatment for CIN2. Gynecol Oncol. 2018 Nov;151(2):229-234. doi: 10.1016/j.ygyno.2018.08.033. Epub 2018 Sep 6. No abstract available. PMID 30197061
- [Result] Pieralli A, Bianchi C, Auzzi N, Fallani MG, Bussani C, Fambrini M, Cariti G, Scarselli G, Petraglia F, Ghelardi A. Indication of prophylactic vaccines as a tool for secondary prevention in HPV-linked disease. Arch Gynecol Obstet. 2018 Dec;298(6):1205-1210. doi: 10.1007/s00404-018-4926-y. Epub 2018 Oct 10. PMID 30306310
- [Result] Velentzis LS, Brotherton JML, Canfell K. Recurrent disease after treatment for cervical pre-cancer: determining whether prophylactic HPV vaccination could play a role in prevention of secondary lesions. Climacteric. 2019 Dec;22(6):596-602. doi: 10.1080/13697137.2019.1600500. Epub 2019 Apr 29. PMID 31030590
- [Result] Paavonen J, Naud P, Salmeron J, Wheeler CM, Chow SN, Apter D, Kitchener H, Castellsague X, Teixeira JC, Skinner SR, Hedrick J, Jaisamrarn U, Limson G, Garland S, Szarewski A, Romanowski B, Aoki FY, Schwarz TF, Poppe WA, Bosch FX, Jenkins D, Hardt K, Zahaf T, Descamps D, Struyf F, Lehtinen M, Dubin G; HPV PATRICIA Study Group. Efficacy of human papillomavirus (HPV)-16/18 AS04-adjuvanted vaccine against cervical infection and precancer caused by oncogenic HPV types (PATRICIA): final analysis of a double-blind, randomised study in young women. Lancet. 2009 Jul 25;374(9686):301-14. doi: 10.1016/S0140-6736(09)61248-4. Epub 2009 Jul 6. PMID 19586656